CLINICAL TRIAL: NCT04163952
Title: A Phase 1 Study of Talimogene Laherparepvec and Panitumumab in Patients With Locally Advanced Squamous Cell Carcinoma of the Skin (SCCS)
Brief Title: Talimogene Laherparepvec and Panitumumab for the Treatment of Locally Advanced or Metastatic Squamous Cell Carcinoma of the Skin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, CINJRegulatory, Principal Investigator is deceased - Professor and Chief of Melanoma and Soft Tissue Sarcoma, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018002628; NCI-2019-06083 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2018002628; 091804 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-11-15 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Skin Squamous Cell Carcinoma; Metastatic Skin Squamous Cell Carcinoma; Recurrent Skin Squamous Cell Carcinoma
MeSH Terms: interventions — Panitumumab; talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talimogene laherparepvec, panitumumab) (Experimental): Patients receive talimogene laherparepvec IM on day 1. Patients then receive talimogene laherparepvec IM and panitumumab IV over 30-90 minutes on day 22. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive up to 3 additional cycles of treatment per physician discretion.
  Interventions: Biological: Panitumumab; Biological: Talimogene Laherparepvec

INTERVENTIONS:
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
Biological: Talimogene Laherparepvec — Given IM
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC

SUMMARY:
This phase I trial studies the side effects and how well talimogene laherparepvec and panitumumab work in treating patients with squamous cell carcinoma of the skin that has spread to nearby tissues or lymph nodes (locally advanced) or other places in the body (metastatic). Talimogene laherparepvec is a type of vaccine made from a gene-modified virus that may help the body build an effective immune response to kill tumor cells. Immunotherapy with monoclonal antibodies, such as panitumumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving talimogene laherparepvec and panitumumab may work better in treating patients with squamous cell carcinoma of the skin compared to panitumumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of the combined treatment of talimogene laherparepvec and panitumumab.

II. To determine the preliminary efficacy of the combined treatment of talimogene laherparepvec and panitumumab, in comparison to single-agent panitumumab by historical control.

SECONDARY OBJECTIVES:

I. To assess the clinical efficacy of panitumumab in combination with intratumoral talimogene laherparepvec in terms of immune-related progression-free survival (irPFS) at 12 months, progression-free survival (PFS) hazard ratio, overall response rate (ORR), 1-year survival, overall survival (OS) and time to resectability.

II. To measure the pathologic complete response rate to panitumumab combined with talimogene laherparepvec.

III. Assess the response of injected and non-injected tumor deposits after panitumumab and talimogene laherparepvec.

IV. Assess the time to initial response. V. Assess the durable response rate.

VI. To analyze the following molecular correlates with response to therapy to confirm mechanism of action, and identify potential future targeted strategies and biomarkers of response:

VIa. Mutation load in tumor tissue by next generation sequencing. VIb. Deoxyribonucleic acid (DNA) mutation signature in tumor tissue pre- and post-therapy by next generation sequencing.

VIc. Messenger ribonucleic acid (mRNA) signature in tumor tissue pre-and post-therapy by Nanostring technology.

VId. Immune cell populations and immune profile in pre- and post-therapy tumor tissue and peripheral blood by flow cytometry and immunohistochemistry (IHC).

OUTLINE:

Patients receive talimogene laherparepvec intratumorally (IM) on day 1. Patients then receive talimogene laherparepvec IM and panitumumab intravenously (IV) over 30-90 minutes on day 22. Treatment repeats every 2 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive up to 3 additional cycles of treatment per physician discretion.

After completion of study treatment, patients are followed up at 30 days and then every 2 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the skin (SCCS) that is a) locally advanced or metastatic for which curative surgery or radiation would be difficult or impossible, or b) recurrent after initial surgery, chemotherapy, or radiation therapy, or c) considered to have aggressive features including the following: tumors 2 cm or more, tumors invading deep tissues such as muscle, cartilage or bone; tumors showing perineural invasion, and/or tumors metastatic to loco-regional lymph nodes. Patients may have had prior surgical interventions or been treated with investigational agents with residual or recurrent disease
* Tumor suitable for direct or ultrasound-guided injection defined as at least one cutaneous, subcutaneous, or nodal lesion, or aggregate of lesions, >= 10 mm in diameter
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* No prior treatment with panitumumab or talimogene laherparepvec for advanced disease
* Prior surgery or radiation is allowed if there is documented progression in the radiated/resected area or elsewhere by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version (v) 1.1
* Measurable disease by RECIST criteria v 1.1
* Patients with a history of hematologic or solid organ transplant will be considered if they do not require high dose steroids or high dose immunosupressants for disease control or control of transplant rejection, and have adequate hematologic, renal, and hepatic function as specified below. Current medications must be reviewed with transplant pharmacy team to exclude potentially serious interactions and case discussed with the study principal investigator (PI)
* Second primary malignancy only if treatment would interfere with the patient?s participation in this trial in the opinion of the treating physician. Clear exceptions are 1) patient had a second primary malignancy but has been treated and disease free for at least 3 years, 2) in situ carcinoma (e.g., in situ carcinoma of the cervix) and, 3) additional skin cancers that have been definitively treated by surgery and/or radiation. Patients with chronic lymphocytic leukemia will be allowed if their blood counts are within acceptable hematologic parameters and if they are not currently requiring cytotoxic or biologic anticancer treatment (supportive treatment such as intravenous immunoglobulin [IVIG] is permitted)
* Patients with autoimmune disorders will be considered if they do not require high dose steroids or other immunosuppressants for disease control. Prednisone in daily doses up to 10 mg and inhaled steroids are acceptable
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count >= 100,000/mm^2
* Hemoglobin >= 9 g/dL
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN); if patient has conditions of congenital hyperbilirubinemia, then patient must have isolated hyperbilirubinemia (e.g., no other liver function test abnormalities) with maximum bilirubin < 2 x institutional ULN
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 x institutional ULN in absence of liver metastases; =< 5 x ULN in presence of liver metastases
* Alkaline phosphatase < 2.5 x institutional ULN
* Creatinine < 1.5 x institutional ULN or calculated creatinine clearance >= 60 mL/min as estimated using the Cockcroft-Gault formula

Exclusion Criteria:

* Pregnant women. Women of childbearing age must be willing to undergo a pregnancy test prior to therapy and to use adequate contraception (e.g., hormonal or barrier method of contraception or abstinence) for the duration of the study and 6 months thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Menopausal status will be defined as one or more of successful hysterectomy, bilateral tubal ligation or bilateral oophorectomy, amenorrhea >= 12 consecutive months without another cause, or a documented serum follicle stimulating hormone (FSH) >= 35 mIU/mL
* Tumor not suitable for direct or ultrasound-guided injection
* Prior treatment with talimogene laherparepvec for advanced disease
* Patients with active, uncontrolled infections including active herpetic infections or chronic herpetic infections requiring anti-viral therapy (e.g., acyclovir)
* Patients without adequate organ function as documented above
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to panitumumab, talimogene laherparepvec or other agents used in the study
* History of interstitial pneumonitis, pulmonary fibrosis, or evidence of interstitial pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Berger, MD, FACS, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - New York University Langone Medical Center, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - Duke University Medical Center - Duke Cancer Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Talimogene Laherparepvec, Panitumumab): Participants receive Talimogene Laherparepvec IM on day one. Participants then receive Talimogene Laherparepvec IM and panitumumab IV over 30-90 minutes on day 22. Treatment repeats every two weeks for up to three cycles in the absence of disease progression or unacceptable toxicity. Participants may receive up to three additional cycles of treatment per physician discretion.
  Panitumumab: Given IV
  Talimogene Laherparepvec: Given IM
Period: Overall Study
Arm/Group | Treatment (Talimogene Laherparepvec, Panitumumab)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Talimogene Laherparepvec, Panitumumab)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by CTCAE v4.0
Description: Number of participants who experience adverse effects greater than or equal to a grade three as defined by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Grade 1-4, with 4 being the most severe.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Talimogene Laherparepvec, Panitumumab)
Number analyzed (Participants) | 5
Participants | 2

2. Primary Outcome: Response Rate to Panitumumab as Measured by Evaluation of the Criteria in Solid Tumors (RECIST) 1.1.
Description: Response will be evaluated by using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Changes in the largest diameter (unidimensional measurement)of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used for tumor measurements.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: Best Overall Response Rate (ORR) of Participants From Start to Progression of Disease
Description: Best response on treatment was based on RECIST 1.1 criteria. Complete response (CR) is complete disappearance of all targeted lesions. Partial response (PR) is at least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference baseline sum. LD Progressive disease (PD) is at least 20% increase in the sum of the longest diameter of the targeted lesions, taking as reference the smallest sum recorded in treatment PD for the evaluation of non-targeted lesions is the appearance of one or more new lesions and or progression of non-targeted lesions. Stable disease is defined as any condition not meet above criteria. The response rate of the drug will be assessed according to the decision rule based on Simons two-stage design.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Durable Response Rate Based on Simons Two-stage Design
Description: Will be defined as the percent of participants with complete response or partial response maintained continuously for a minimum of six months. The response rate of the drug will be assessed according to the decision rule based on Simons two-stage design.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Duration of Response Based on Simons Two-stage Design
Description: The response rate of the drug will be assessed according to the decision rule based on Simon?s two-stage design.
Time Frame: Time from initial response until document progression up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Progression-free Survival (PFS) to Assess Participants Progressive Free-survival
Description: The estimate of PFS will be performed by the Kaplan-Meier product limit model.>valuated by RECIST 1.1.
Time Frame: From date of enrollment to the date of death or progression, whichever occurred earlier assessed up to 2 years
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Change in Overall Survival (OS) Measured by the Kaplan-Meier
Description: The estimate of OS will be performed by the Kaplan-Meier product limit model.
Time Frame: From date of enrollment to the date of death or date last known alive, whichever comes first, assessed up to assessed up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Mutation Load in Tumor Tissue Measured by Next Generation Sequencing
Description: Next generation sequencing (NGS) is a massively parallel sequencing technology that offers ultra-high throughput, scalability, and speed. The technology is used to determine the order of nucleotides in entire genomes or targeted regions of DNA or RNA, and has the ability to detect variants at lower allele frequencies. With response to therapy and but the actual knowledge of the genetic basis of participants disease.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Deoxyribonucleic Acid Mutation Signature in Tumor Tissue
Description: Will be analyzed by next generation sequencing with response to therapy.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Messenger Ribonucleic Acid Signature in Tumor Tissue Measured by Nanostring Technology
Description: Nanostring is an amplification-free technology that measures nucleic acid content by counting molecules directly. NanoString provides several pre-made gene expression panels that examine up to 770 genes at once and custom CodeSets for up to 800 targets. With response to therapy and descriptive statistics applied.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-02

11. Secondary Outcome: Immune Cell Populations in Tumor Tissue
Description: Will be analyzed by flow cytometry with response to therapy.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Immune Cell Populations Peripheral Blood as Measured by Flow Cytometry
Description: Cytometry, in its purest form, is the measurement of cell characteristics. Flow cytometry can identify the type of cells in a blood or bone marrow sample, including the types of cancer cells. It detects types of cancer cells based on either the presence or the absence of certain protein markers (antigens) on a cell's surface. This technique allows researchers to get highly specific information about individual cells. Flow cytometry will be used, with response to therapy and descriptive statistics applied.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Expression of Cytokines in Tumor Tissue
Description: Will be analyzed by flow cytometry, any suspended particle or cell from 0.2-150 micrometers in size, is suitable for analysis.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: Expression of Cytokines in Peripheral Blood
Description: Will be analyzed by flow cytometry, any suspended particle or cell from 0.2-150 micrometers in size is suitable for analysis, with response to therapy.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Pathologic Complete Response Rate
Description: Pathologic complete response (pCR) was defined as percent necrosis of the surgical specimen greater than or equal to 90% .Pathologic complete response (pCR) is a surrogate endpoint to demonstrate the study drug's efficacy.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Time to Resectability
Description: A resectable tumor is one in which there is no technical barrier to surgical excision. Able to be removed by surgery.
Time Frame: Up to two years
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: From date of enrollment to the date of death or progression, whichever occurred earlier assessed up to two years.
Arm/Group | Treatment (Talimogene Laherparepvec, Panitumumab)
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Talimogene Laherparepvec, Panitumumab) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Talimogene Laherparepvec, Panitumumab) (N=5)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (10)
Fever (General disorders) | 2 (6)
Chills (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT04163952/Prot_SAP_002.pdf
  • Informed Consent Form: ICF 1 (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT04163952/ICF_000.pdf